CLINICAL TRIAL: NCT06087224
Title: The TELENEO Trial: A Multicenter Trial of Telemedicine for Advanced Neonatal Resuscitations in Community Hospitals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jennifer L. Fang, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-005502; R01HD112327 (NIH)
Record Dates: First submitted 2023-10-12; First posted 2023-10-17 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Death; Neonatal; Morbidity;Newborn
Keywords: Telemedicine; Newborn; Resuscitation
MeSH Terms: conditions — Perinatal Death

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teleneonatology group (Experimental): Study eligible neonates cared for by the community hospital team with telemedicine consultation by a neonatologist from the regional neonatal intensive care unit (NICU).
  Interventions: Other: Teleneonatology
- Control group (No Intervention): Study eligible neonates cared for by the community hospital team per the site's usual practice of care.

INTERVENTIONS:
Other: Teleneonatology — Real-time, two way, audio-video telemedicine connection between the neonatologist located in the regional neonatal intensive care unit (NICU) and the physician located at the community hospital.
  Arms: Teleneonatology group

SUMMARY:
The purpose of this study is to evaluate the impact of real-time audio-video telemedicine consults with a neonatologist (termed teleneonatology) on the early health outcomes of at-risk neonates delivered in community hospitals.

DETAILED DESCRIPTION:
This prospective, multicenter trial will use a stepped wedge cluster randomized study design to evaluate the impact of real-time audio-video telemedicine consults with a neonatologist (termed "teleneonatology") on the risk of early mortality, early morbidity, and delivery room care for at-risk neonates delivered in community hospitals.

ELIGIBILITY:
Inclusion Criteria:

GROUP 1: Community hospital clinicians

To be eligible to participate in this study, an individual must meet all of the following criteria:

1. A clinician who attends newborn resuscitations at a participating community hospital spoke site.
2. Provision of informed oral consent prior to any mandatory study specific procedures and analyses.

GROUP 2: At-risk outborn neonates To be eligible for this study, a neonate born in a participating community hospital spoke site must meet *at least one* of the following inclusion criteria

1. Preterm birth at less than 32 weeks' gestation at delivery; OR
2. Need for advanced resuscitation defined as:

   1. positive pressure ventilation (PPV) initiated soon after birth and continued for at least 10 minutes; OR
   2. placement of an alternative airway (endotracheal tube or laryngeal mask) to provide PPV; OR
   3. chest compressions.

Exclusion Criteria:

GROUP 1: Community hospital clinicians None

GROUP 2: At-risk outborn neonates

A neonate born in a participating community hospital spoke site who meets any of the following criteria will be excluded from the study:

1. Birth outside of the hospital birthing center.
2. Neonatal transport team present at time of birth and providing resuscitative care.
3. Severe congenital anomaly necessitating intensive care or surgery in the first two weeks of life.
4. Plan for comfort care (non-resuscitation) following delivery.
5. In-person neonatology-trained physician present for the resuscitation.

Min Age: 0 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 947 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2029-02-07 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
7-day mortality rate | 7 days
  Percentage of neonates classified as dying within 7 days, defined as death on or before 23:59 on the seventh completed day of life.

SECONDARY OUTCOMES:
Early neonatal morbidity within the first 7 days | 7 days
  Percentage of neonates classified as having early neonatal morbidity, defined as diagnosed with definite pneumothorax on chest imaging, severe intracranial hemorrhage on brain imaging (grade 3 or 4 intraventricular hemorrhage per Papile classification or cerebellar hemorrhage), or seizures on electroencephalogram in the first seven days of life
Composite outcome of early mortality and morbidity | 7 days
  Percentage of neonates classified as having early neonatal mortality or morbidity, defined as dying or diagnosed with definite pneumothorax on chest imaging, severe intracranial hemorrhage on brain imaging, or seizures on electroencephalogram in the first seven days of life.
Highest level of resuscitation received in the delivery room | First hour of life
  The highest level of delivery room resuscitation during the first hour of life, on a scale of 1-6, corresponding to routine care; oxygen and/or continuous positive airway pressure (CPAP); positive pressure ventilation (PPV); advanced airway placement (endotracheal tube or laryngeal mask); chest compressions; or epinephrine administration, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Fang, MD, Principal Investigator — Mayo Clinic; Bart M Demaerschalk, MD, Principal Investigator — Mayo Clinic; Meegan G Van Straaten, MSPH, Study Director — Mayo Clinic
Locations (36):
- United States (21):
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Bartlett Regional Hospital, Juneau, Alaska
  - PeaceHealth Ketchikan Medical Center, Ketchikan, Alaska
  - Mayo Clinic Arizona, Pheonix, Arizona
  - Mayo Clinic Minnesota, Rochester, Minnesota
  - Chickasaw Nation Medical Center, Ada, Oklahoma
  - Jackson County Memorial Hospital, Altus, Oklahoma
  - Great Plains Regional Medical Center, Elk City, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Island Health, Anacortes, Washington
  - Providence Regional Medical Center Everett, Everett, Washington
  - Olympic Medical Center, Port Angeles, Washington
  - Seattle Children's Hospital, Seattle, Washington
  - University of Washington, Seattle, Washington
  - Central Washington Health Services Association d/b/a Confluence Health, Wenatchee, Washington
  - Prairie Ridge Health, Columbus, Wisconsin
  - Fort HealthCare, Fort Atkinson, Wisconsin
  - University of Wisconsin-Madison, Madison, Wisconsin
  - Sauk Prairie Healthcare, Prairie du Sac, Wisconsin
  - Reedsburg Area Medical Center, Reedsburg, Wisconsin
  - Watertown Regional Medical Center, Watertown, Wisconsin
- Canada (15):
  - Stevenson Memorial Hospital, Alliston, Ontario
  - William Osler Health System - Brampton Civic Hospital, Brampton, Ontario
  - Michael Garron Hospital, East York, Ontario
  - William Osler Health System - Etobicoke General Hospital, Etobicoke, Ontario
  - Trillium Health Partners - Credit Valley Health, Mississauga, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Orillia Soldiers Memorial Hospital, Orillia, Ontario
  - Scarborough Health Network - Centenary Hospital, Scarborough Village, Ontario
  - Scarborough Health Network - General Hospital, Scarborough Village, Ontario
  - North York General Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Unity Health - St. Joseph's Health Centre, Toronto, Ontario
  - Mackenzie Health - Cortellucci Vaughan Hospital, Vaughan, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fang JL, Umoren R, Whyte H, Limjoco J, Makkar A, Yankanah R, McCoy M, Lo MD, Colby CE, Herrin J, Jacobson RM, Demaerschalk BM. Provider Perspectives on the Acceptability, Appropriateness, and Feasibility of Teleneonatology. Am J Perinatol. 2023 Oct;40(14):1521-1528. doi: 10.1055/a-1656-6363. Epub 2021 Sep 28. PMID 34583392
- [Background] Fang JL, Whyte H, Umoren R, Limjoco J, Makkar A, Yankanah R, McCoy M, Lo MD, Herrin J, Demaerschalk BM. Accuracy of Simulated Research Tasks by Community Hospitals Participating in a Multicenter Telemedicine Trial. Telemed J E Health. 2022 Oct;28(10):1489-1495. doi: 10.1089/tmj.2021.0574. Epub 2022 Feb 15. PMID 35167373
- [Background] Fang JL, Umoren RA, Whyte H, Limjoco J, Makkar A, Behl S, Lo MD, White L, Culjat M, Taylor JS, Kathuria S, Webb MO, Schad T, Shafranski S, Yankanah R, Herrin J, Demaerschalk BM. Evaluating the feasibility of a multicenter teleneonatology clinical effectiveness trial. Pediatr Res. 2023 Oct;94(4):1555-1561. doi: 10.1038/s41390-023-02659-2. Epub 2023 May 19. PMID 37208433
- See also: Mayo Clinic Clinical Trials — https://www.mayoclinic.org/teleneonatology-program/clinical-trials